CLINICAL TRIAL: NCT04084093
Title: Evaluating the Use of a Concentrated Surfactant Gel in Burn Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will be redesigned.
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2018-DIV31-011
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2019-09

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: This device is helps in the creation of an optimal moist wound healing environment that aids in protecting healthy tissues and provides an environment conductive to autolytic debridement. The device is 100% water-soluble, biocompatible, and non-ionic. The dressing is a surfactant based gel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surfactant Gel (Experimental)
  Interventions: Device: Surfactant Gel

INTERVENTIONS:
Device: Surfactant Gel — This device is helps in the creation of an optimal moist wound healing environment that aids in protecting healthy tissues and provides an environment conductive to autolytic debridement. The device is 100% water-soluble, biocompatible, and non-ionic. The dressing is a surfactant based gel.

SUMMARY:
This will be an observational study evaluating subject's perception of pain to dressing changes during removal and application of a surfactant gel. Wound healing will also be monitored. Anxiety before dressing change will be measured using a burn specific pain anxiety scale. Study intervention will include cleansing the wound per the facility's standard of care, followed by applying the investigational product on the wound. This will be followed by placing an appropriate secondary dressing.

ELIGIBILITY:
Inclusion Criteria:

* Subject should be an inpatient, per the Two-Midnight rule at the time of study initiation.
* At the time of subject's admission in the hospital, duration of his or her burn wound should be < or equal to 24 hours.
* Subject who has a partial thickness burn wound, or an indeterminate burn wound, or who has both these characteristics in the same wound, as determined by the site Principal Investigator.
* Subject's wound included in this study, does not require any surgical intervention.
* Subject is able and willing to comply with requirements of this trial protocol.
* Voluntarily signed informed consent obtained before any trial-related procedures are performed.
* Subject must be able to communicate effectively with study personnel.
* Subject has burn total body surface area (TBSA) between 1-20%.

Exclusion Criteria:

* Subjects with electrical or radiation burns.
* Subjects who are pregnant, nursing or planning to become pregnant during the course of the study.
* Subjects who have known allergies to any ingredients in the dressings used in the study.
* Subjects taking opiates during the study duration.
* Subjects with an active diagnosis of substance use disorder within the past six months.
* Subjects with previously diagnosed issues with pain perception, including conditions such as peripheral neuropathy, if they will preclude accurate assessment of primary and secondary endpoints.
* Subjects with an active infection prior to enrollment.
* Subject has previous or current systemic disease(s) which, in the judgement of the investigator, is likely to interfere with treatment. Subjects with well-controlled diabetes mellitus (HbA1C<8.5) shall be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Self-reported evaluation of subject pain perception during dressing changes using a numerical pain scale. | Baseline to Day 30
  The numerical pain scale will be from 0 to 10 with 0 being no pain at all and 10 being the worst pain ever possible. This is the numeric rating scale.

SECONDARY OUTCOMES:
Measure percent change in epithelium as recorded by the clinician. | Baseline to Day 30
Measure percent change in necrotic tissue in the wound bed | Baseline to Day 30
Measure change in wound size | Baseline to Day 30
Measure anxiety using a burn specific anxiety scale | Baseline to Day 30
  A burn-specific pain anxiety scale will be used to measure level of anxiety. Items will be scored on a 100mm visual analog line with two reference points, 0 and 100. These reference points will also be identified by expressions "not at all" and "the worst imaginable way". Subjects will be requested to scale the strength of their feelings relative to two reference points.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: No